CLINICAL TRIAL: NCT02631330
Title: Effect on Falls Reduction of a Multimodal Intervention in Frail and Pre-frail Elderly Community-dwelling People in Madeira Island (Portugal) and Valencia (Spain)
Brief Title: Effect on Falls Reduction of a Multimodal Intervention in Frail and Pre-frail Elderly Community-dwelling People
Acronym: FAREMAVA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de la Ribera (Other)
Responsible Party: Principal Investigator, Francisco Jose Tarazona-Santabalbina, MD, PhD, Consultant in Geriatric Medicine Hospital Universitario de la Ribera. Associated Professor Universidad Católica de Valencia San Vicente Mártir, Hospital de la Ribera
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FAREMAVA2015
Record Dates: First submitted 2015-12-03; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Accidental Falls
Keywords: Geriatric Assessment; Physical Education and Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Falls prevention group (Experimental): Intervention group that will receive a monthly talk (individual or collective) of 30 minutes on the advantages of having a free fall hazards environment and multiple physical exercise component: balance,muscle strength and aerobic capacity and risk polypharmacy and abuse of drugs, especially benzodiazepines). In the same monthly meeting, subjects will be train "Multicomponent physical activity" program during 60 minutes. 15 minutes of gait and balance training; 15 minutes of endurance training; 30 minutes of aerobic training according Training Intervention in a Controlled Population of Frail Elderly (EMTIFE) study NCT02331459
  Interventions: Other: Multicomponent physical activity
- Control group (No Intervention): Subjects will receive the same information provided at the beginning to Falls prevention group. They will not receive further information during the follow-up period.

INTERVENTIONS:
Other: Multicomponent physical activity — Balance, muscle strength and aerobic capacity will be increased in intensity according Training Intervention in a Controlled Population of Frail Elderly (EMTIFE) study NCT02331459
  Arms: Falls prevention group

SUMMARY:
Practice guidelines in caring for the geriatric population recommend performing an annual screening of falls . However, one of the problems that interfere with fall prevention programs is the lack of importance accorded to health professionals to falls. This lack of awareness of the risks faced by the associated geriatric population falls generates reluctance to adherence to a fall prevention program . At European level there are the same gaps in knowledge about the real effectiveness and efficiency of fall prevention programs .

HYPOTHESIS: The implementation of a multicomponent fall prevention program in frail and pre-frail elderly community-dwelling people reduce the incidence of falls.

OBJECTIVES

General:

• To determine the efficacy of a comprehensive program to prevent falls in the community.

Specific:

* Knowing whether reducing the incidence of falls implies a reduction in visits to primary care, emergency department or hospital staying.
* Knowing the adhesion, through indirect measures, to the intervention program.
* Knowing the nutritional, functional, cognitive, social, anthropometric, respiratory and clinical profile, including falls, of the sample.

MATERIAL AND METHODS

Study design:

Multicenter community intervention study, longitudinal, prospective, randomized, and experimental.

Through intervention by nurses in primary care education of subjects over 70 years it is to know the effectiveness of a comprehensive program of falls prevention.

It will proceed to recruit older than or equal to 70 years subjects, who meet frailty criteria age, belonging to the areas of Madeira Island (Portugal) and La Ribera County (Valéncia, Spain) .

DETAILED DESCRIPTION:
INTRODUCTION The World Health Organization (WHO) defines fall as a result of any event precipitating the patient down, involuntarily .

Along with instability and gait disturbances, falls are one of the great geriatric syndromes and are the second cause of death worldwide by unintentional injuries.

In the field of public health, falls in the elderly are considered a major biopsychosocial problem due to medical, psychological, social and family and economic consequences. It is estimated that in 2020 the cost generated to the social and health care by falls will be about 30,000 million euros. This is because about 20% of falls require medical attention, with approximately 10% of consultations in emergency services and 6% of urgent hospitalization in the elderly .

Mortality in elderly people as a result of falls is nearly 40,000 deaths annually in Europe, obtaining in Spain a mortality rate 15 . It also has a high morbidity, as declines are directly related to decreased mobility and ability to perform basic activities of daily living, raising fears of a new fall and thus favoring the loss of one's safety same. Thus the dependence on a caregiver or institutionalization in a home increases, in turn, the family, social and economic impact.

Falls in the elderly, unlike the adult, are the result of the adaptive imbalance of the person from the environment. The clinician relativizes this problem by attributing the fall to the normal aging process and ignore its potential consequences: injury, disability, institutionalization and even death in this population. For this reason, falls are considered a factor of frailty in the elderly .

The performance of health workers to a fall in the elderly patient should consist of the realization of the following measures :

* Conduct a comprehensive assessment of elderly: biomedical, functional, social, mental and psycho-sphere.
* Identify intrinsic, extrinsic risk factors and circumstances of the fall.
* Estimate early physical, psychological and socio-economic consequences.
* Prevention of falls at primary, secondary and tertiary levels. Frailty is a pathophysiological syndrome characterized by decreased functional reserve which is mainly linked to the loss of muscle mass or sarcopenia. This is caused by the decline in physical activity, associated in turn with poor health habits, cardiovascular risk factors and various chronic diseases. The consequences in the elderly affect multiple systems , causing greater vulnerability to external agents and increasing the risk: disability, hospitalization, institutionalization and death . The prevalence of frailty in subjects over 65 years is between 7 and 16.3% , increasing every decade from this age .

The diagnostic criteria for fragility, described by Linda Fried, include the assessment of functional aspects as the gait assessment, exhaustion or strength of palmar pressure with weight loss and energy consumption associated with physical activity . Since therapeutic perspective, one of the best ways to reverse the frailty is the physical exercise. Several articles have described heterogeneous effects on physical interventions in elderly frailty people , ranging from isolated programs of aerobic, anaerobic or balance to different combinations of the same training. A multicomponent exercise program increased muscle strength, improve cardiorespiratory fitness and balance11. Exercise programs have observed improvement in symptoms of depression in elderly patients10 up to 3 months after completion of the program . This benefit may be due to increased central monoamine activity and increased secretion of beta-endorphin. Similarly, it has been linked exercise programs with improvement in various cognitive domains, especially in executive functions. A 2003 meta-analysis indicates that the combined program of aerobic and anaerobic exercise have a better outcome on cognitive status than those designed with only aerobic programs.

STUDY JUSTIFICATION Nearly six million Spanish people are older than 70 years, 12.64% of the Spanish population is elderly. The first study in Spain on falls in the elderly was conducted in 1985 and from then until now, it has encouraged the investigation.

Practice guidelines in caring for the geriatric population recommend performing an annual screening of falls . Moreover, they suggest to advice the elderly on possible risk factors associated. However, one of the problems that interfere with fall prevention programs is the lack of importance accorded to health professionals to falls. This lack of awareness of the risks faced by the associated geriatric population falls generates reluctance to adherence to a fall prevention program .

At European level there are the same gaps in knowledge about the real effectiveness and efficiency of fall prevention programs .

Add the practice of physical activity in nursing interventions, under the environment of the community, have shown a reduction in the use of emergency services at relatively short intervals, probably due to improved continuity of care .

The Hunter study showed that a training program low-level resistance (twice a week) is associated with a decrease in the progression of functional limitations within 6 months.

Physical activity associated with an interdisciplinary approach improves overall assessment of the frail elderly population on the functional, psychological, cognitive, clinical and social part , , , .

It is necessary to create an interdisciplinary team in daily clinical practice in frail patients to perform adequately the full recognition of these patients with the following characteristics:

* Shared management between nursing and primary care.
* Support staff (nurses, social workers) with specialized training in gerontology.
* Audit of the home and technical devices needs.
* Regular team meetings to evaluate changes.
* Establishment of communication with community resources to incremental improvements in the home, health promotion and support to caregivers.

HYPOTHESIS The implementation of a multicomponent fall prevention program in frail and pre-frail elderly community-dwelling people reduce the incidence of falls.

OBJECTIVES

General:

• To determine the efficacy of a comprehensive program to prevent falls in the community.

Specific:

* Knowing whether reducing the incidence of falls implies a reduction in visits to primary care, emergency department or hospital staying.
* Knowing the adhesion, through indirect measures, to the intervention program.
* Knowing the nutritional, functional, cognitive, social, anthropometric, respiratory and clinical profile, including falls, of the sample.

MATERIAL AND METHODS

Study design:

Multicenter community intervention study, longitudinal, prospective, randomized, and experimental.

Through intervention by nurses in primary care education of subjects over 70 years it is to know the effectiveness of a comprehensive program of falls prevention.

ELIGIBILITY:
Inclusion Criteria:

* Women and men with older than or equal to 70 years old.
* Independent ambulation (may have technical aids but not someone else).
* Usual residence in the areas of health described.
* Linda Fried's Criteria of pre-frailty or frailty.

Exclusion Criteria:

* Patients with life expectancy of less than six months.
* Institutionalized patients.
* Patients with severe hearing or visual deficits.
* Patients with contraindication in physical exercise.
* Patients with serious psychiatric illness or moderate or severe cognitive impairment.
* Patients who refuse to sign the informed consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Falls incidence change | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Number of falls observed during the follow up period

SECONDARY OUTCOMES:
Primary care and emergency department visits related with falls | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Number of visits related with falls observed during the follow up period in primary attention services, emergency departments and hospital admissions
Changes in nutritional status | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Change in nutritional parameters (MNA score) between groups during follow up period
Changes in functional status | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Changes in the following variable during follow up period: SHORT PHYSICAL PERFORMANCE BATTERY,
Changes in cognitive status | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Changes in the following variable during follow up period: MMSE
Changes in anthropometric measures | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Changes in the following variable during follow up period: BMI
Changes in respiratory function | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Changes in the following variables during follow up period
  : FVC, FEV1, FEV1/FVC, MEF25/75, FEV25, FEV50, FEV75, PEF, MIP (Maximal inspiratory pressure) (ELKA-PM15)®, MEP (Maximal espiratory pressure) (ELKA-PM15)®
Changes in daily living autonomy | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Changes in the following variables during follow up period
  : BARTHEL SCALE LAWTON SCALE
Changes in quality of life | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Changes in the following variables during follow up period
  :EUROQOL-5D
Changes in mood state | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Changes in the following variable during follow up period
  :Yesavage Geriatric Depression Scale.
Changes in clinical aspects | day 0, day 90, day 180, day 270 and day 365 (plus or minus 5 days)
  Changes in the following variable during follow up period
  : Hospital admissions rate related with falls

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Tarazona-Santabalbina, MD,PhD, Principal Investigator — Hospital Universitario de la Ribera
Locations (1):
- Hospital Universitario de la Ribera, Alzira, Valéncia, Spain

REFERENCES:
- [Background] Cadore EL, Rodriguez-Manas L, Sinclair A, Izquierdo M. Effects of different exercise interventions on risk of falls, gait ability, and balance in physically frail older adults: a systematic review. Rejuvenation Res. 2013 Apr;16(2):105-14. doi: 10.1089/rej.2012.1397. PMID 23327448
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Porter Starr KN, McDonald SR, Bales CW. Obesity and physical frailty in older adults: a scoping review of lifestyle intervention trials. J Am Med Dir Assoc. 2014 Apr;15(4):240-50. doi: 10.1016/j.jamda.2013.11.008. Epub 2014 Jan 17. PMID 24445063
- [Background] Vivrette RL, Rubenstein LZ, Martin JL, Josephson KR, Kramer BJ. Development of a fall-risk self-assessment for community-dwelling seniors. J Aging Phys Act. 2011 Jan;19(1):16-29. doi: 10.1123/japa.19.1.16. PMID 21285473
- [Background] Theou O, Stathokostas L, Roland KP, Jakobi JM, Patterson C, Vandervoort AA, Jones GR. The effectiveness of exercise interventions for the management of frailty: a systematic review. J Aging Res. 2011 Apr 4;2011:569194. doi: 10.4061/2011/569194. PMID 21584244